CLINICAL TRIAL: NCT01501838
Title: Pulmonary Hypertension Institutional Registry at Hospital Italiano de Buenos Aires
Acronym: PH-HIBA
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Ignacio M Bluro, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 1487
Record Dates: First submitted 2011-06-16; First posted 2011-12-29 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Hypertension, Pulmonary Arterial
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a registry of patients with Pulmonary Hypertension who received medical care in the Hospital Italiano of Buenos Aires.

DETAILED DESCRIPTION:
The Institutional Registry of Pulmonary Hypertension includes patients prospectively with incident pulmonary hypertension type I. It also includes prevalent cases from our HMO who had diagnosis prior the beginning of the registry.

ELIGIBILITY:
* Inclusion Criteria:

  1. Diagnosed with PAH WHO group 1 (2022 ESC/ESR guidelines criteria) as the presence of a mean pulmonary artery pressure (mPAP) greater than 20 mmHg at rest with pulmonary arterial wedge pressure (PAWP) >15 mmHg and pulmonary vascular resistance (PVR) >2 WU, according to the 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension.
  2. Included in the institutional registry of PAH of Hospital Italiano de Buenos Aires
  3. Aged ≥18 years at the index date.
* Exclusion Criteria History of lung transplantation surgery previously the baseline period

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who meet inclusion criteria and none of exclusion criteria during the study period are eligible to this study. In the population, the PAH cohort will consist of those incident cases and prevalent cases PAH WHO group 1 aged ≥18 years between January 2017 and December 2030 who attended at Hospital Italiano of Buenos Aires.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Hypertension prevalence | 1 year
  Pulmonary Hypertension prevalence in our community.
Pulmonary Hypertension incidence | 1 year
  Pulmonary Hypertension incidence in our community

SECONDARY OUTCOMES:
Mortality rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio M Bluro, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided